CLINICAL TRIAL: NCT00617110
Title: Effects of Diesel Exhaust Particles on Influenza-induced Nasal Inflammation in Allergic Rhinitics and Non-allergic Individuals
Brief Title: Effects of Diesel Exhaust Followed by Administration of Nasal Spray Flu Vaccine on Individuals With & Without Allergies
Acronym: FLAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH); Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Terry Noah, MD, Professor of Pediatrics, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 07-1064; 2R01ES013611 (NIH)
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Allergic Rhinitis
Keywords: diesel exhaust particles; live attenuated influenza virus vaccine; flu vaccine
MeSH Terms: conditions — Rhinitis, Allergic; Influenza, Human | interventions — FluMist

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- allergic clean air (Sham Comparator): subjects with allergic rhinitis will be exposed to clean air followed by LAIV
  Interventions: Other: live attenuated influenza virus (LAIV) with clean air
- Allergic diesel (Active Comparator): subjects with allergic rhinitis will be exposed to diesel exhaust particles followed by LAIV
  Interventions: Other: LAIV and diesel exhaust particles
- control clean air (Sham Comparator): Healthy control subjects will be exposed to clean air followed by LAIV
  Interventions: Other: live attenuated influenza virus (LAIV) with clean air
- Control diesel (Sham Comparator): Healthy control will be exposed to diesel followed by LAIV
  Interventions: Other: LAIV and diesel exhaust particles

INTERVENTIONS:
Other: live attenuated influenza virus (LAIV) with clean air — Allergic subjects will be exposed to air followed by administration of live attenuated influenza virus
  Other Names: FluMist
  Arms: allergic clean air; control clean air
Other: LAIV and diesel exhaust particles — subjects with allergic rhinitis will be exposed to diesel exhaust particles followed by LAIV
  Other Names: FLuMist
  Arms: Allergic diesel; Control diesel

SUMMARY:
Allergic rhinitis (AR) is a condition that exists when an individual with a specific allergy reacts to that allergen resulting in a runny and/or stuffy nose, postnasal drip, and possible symptoms of sneezing, scratchy throat, itchy nose, ears or throat. When the allergic person is exposed to such an allergen, the body reacts with overproduction of certain chemicals which cause inflammation and subsequent symptoms of AR. These responses are related to the body's hyperreactive response to exposure to an otherwise harmless substance such as dust, ragweed, pollen, cat dander etc.

There are data to suggest that air pollution resulting from diesel exhaust can increase the body's response to airway inflammation caused by virus.

The purpose of this research study is to determine if individuals with AR have increased inflammatory responses to flu virus following exposure to diesel exhaust (DE) vs exposure to clean air compared to how individuals who do not have allergies respond to the same exposure conditions. The hypothesis for this study is that diesel exhaust exacerbates LAIV-induced allergic nasal inflammation, using controlled exposures in AR volunteers compared to non-allergic individuals

DETAILED DESCRIPTION:
Screening day: This visit will occur approximately 2-4 weeks before your exposure day. You will come to the research facility where you will discuss this consent form with the study coordinator and complete the signature areas. Your vital signs (pulse, temperature, BP, oxygenation saturation) will be measured and the following evaluations will be performed:

* For females of child bearing potential, a urine pregnancy test
* Review your medical history and any recent health changes
* Completion of a questionnaire regarding your allergy symptoms
* Collection of spirometric (pulmonary function testing) data will be performed. You must demonstrate normal pulmonary function in order to continue in the study. You will be asked to inhale as deeply as possible, then exhale as rapidly and completely as possible into a mouthpiece which is connected to a computer which measures various lung volumes and which will tell us if your lung function is normal.
* Blood draw from a hand or arm vein to test for HIV and recent influenza exposure, as well as serum markers, T cell stimulation and WBC characterization. The volume of blood will be up to 50 cc (approximately 3 tablespoons).
* A buccal swab will be performed for genotyping which entails rubbing a toothbrush on the inside of your cheeks to loosen the cells followed by repeating the rubbing in the same place with a soft swab (similar to a Q tip® with a longer stick).
* Physical examination by a study physician
* Allergy skin test if this has not been performed during the previous 2 years
* Collection of nasal lavage fluid which will involve spraying some salt water into your nose repeatedly and then blowing your nose into a cup
* Nasal biopsy during which the researcher gently scrapes the inside lining of your nose with a plastic stick

Day 0 (Monday): You will be asked to eat a light breakfast and arrive at the EPA in early to mid morning. You will need to wear comfortable clothes and shoes, and bring a lunch.

* Collection of vital sign measurements and update in medical condition as well as medications taken since the previous visit
* Urine pregnancy test, if applicable
* A telemetry monitor will be placed so that your heart rhythm can be monitored during your chamber exposure. This will include having monitor wires attached to your chest and shoulders with an adhesive pad. The other end of the wires is connected to a box that can be tied to your waste and which will transmit your heart rhythm to a screen so we can observe it
* Spirometry measurements: This test measures the volume of air that can be exhaled and the rate of airflow during exhalation after a maximal inhalation. You will inhale as deeply as possible, then exhale as rapidly and completely as possible into the spirometer. Measurements obtained from each maneuver include the forced vital capacity (FVC), the forced expiratory volume in the first second (FEV1), the maximal mid-expiratory flow rate (FEF 25-75%) and the peak flow (PF). The largest FVC and FEV1, from at least 3 acceptable trials, are selected for analysis; the flow rates are selected from the trial with the largest sum of FVC.
* Nasal lavage
* You will have a 2 hour exposure to either diesel particles or air. The type of exposure you will receive will be randomized, meaning that you will be assigned to the air or diesel exposure group by chance, like flipping a coin. The exposure will be double blind which means that neither you nor the study investigators and staff will know whether you are being exposed to diesel exhaust or air except in the event of any emergency when this information could be revealed. If you are randomized to receive a diesel exposure, the diesel will be generated from an engine mounted on a vehicle located outside of the EPA Human studies Facility (HSF). The diesel exhaust (DE) is then introduced into the exposure chamber after dilution with clean filtered and humidified air by approximately 1/30th to give a chamber concentration of approximately 100 μg/m3. The amount of DE used for exposure in this study would be equivalent to concentrations encountered at busy intersections in large urban areas. DE concentrations proposed are below occupational levels for some truck drivers (generally about 100-300 µg/m3) and 1-2 mg/m3 for some mines. Some areas of heavily trafficked streets in Los Angeles and New York City have had DE levels > 20 µg/m3, and nearby residents could have exposure to these concentrations over several hours. If you are randomized to clean air, you will receive Chapel Hill air which has been filtered to remove ambient air pollutants
* After your exposure you will have additional spirometry testing and return to the medical station where you will be monitored for 3 hours. You will also have time to eat your lunch which we are requesting that you bring with you from home
* Both before and after your exposure, the level of carbon monoxide in your blood will be tested
* Three hours after your exposure is complete, the FluMist® vaccine will be administered by spraying the vaccine once into each nostril. Shortly after that you will be discharged home

Days 1-3 (Tuesday-Thursday). Each day, the following will be obtained:

* Vital signs and update any changes in medical condition
* Nasal lavage

Day 4 (Friday):

* Vital signs and medical update
* Nasal lavage
* Nasal biopsy
* Blood draw - serum markers, WBC characterization. The volume of blood will be up to 50cc (approximately 3 tablespoons)

Day 9 +/- 1 day (one visit sometime between the Tuesday through Thursday after the week you have received the FluMist®):

* Vital signs and health update
* Nasal lavage

Day 21 +/-7 days after the FluMist dose

* Vital signs and health update
* Urine pregnancy test, if applicable
* Blood draw to check your post -vaccine anti-influenza titer, as well as serum markers, T cell stimulation and WBC characterization. The volume of blood will be up to 50 cc (approximately 3 tablespoons)

ELIGIBILITY:
Inclusion Criteria:

1. Normal lung function, defined as (Knudsen 1976/1984 predicted set):

   * FVC of > 75 % of that predicted for gender, ethnicity, age and height
   * FEV1 of > 75 % of that predicted for gender, ethnicity, age and height
   * FEV1/FVC ratio of .70
2. Oxygen saturation of > 94 %
3. Normal blood pressure (Systolic between 140 - 90, Diastolic between 90-60 mm Hg)
4. Symptom Score no greater than 6 (out of a possible 39) for total symptom score
5. On the day of a challenge, body temperature must be no greater than 37.8 degrees, measured orally

Exclusion Criteria:

1. A history of significant chronic illnesses (to include diabetes, autoimmune diseases, immunodeficiency state, known ischemic heart disease, chronic respiratory diseases such as chronic obstructive pulmonary disease or asthma, hypertension)
2. Allergy to any medications which may be used in the course of this study (albuterol, acetaminophen, aspirin or non-steroidal anti-inflammatory agents, corticosteroids)
3. Positive pregnancy test within 48 hours of the time of challenge
4. Medications which may impact the results of the experimental viral infection, interfere with any other medications potentially used in the study (to include nasal or oral corticosteroids, beta adrenergic antagonists, non-steroidal anti-inflammatory agents) or suggest an ongoing illness (such as antibiotics)
5. Acute, non-chronic, medical conditions, including (but not limited to) pneumonia or bronchitis requiring antibiotics, febrile illnesses, flu-like symptoms must be totally resolved symptomatically for 3 weeks
6. Unspecified illnesses, which in the judgment of the investigator increase the risk associated with the experimental LAIV infection, will be a basis for exclusion
7. Use of any inhaled substance (for medical or recreational purposes)
8. Receipt of flu vaccine of any type (injection or nasal spray) during the prior season (2006/2007)
9. Current use of allergy immunotherapy ("allergy shots")

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2008-01; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in IL-13 and ECP in nasal lavage fluids (NLF) compared to pre-virus baseline | 1-21 days post challenge

SECONDARY OUTCOMES:
Duration/quantity of virus shedding | 0-21 days post challenge
Change in inflammatory cells in NLF at specific time points compared to baseline | 0-21 days post challenge
Change in inflammatory cytokines/chemokines and other mediators (PGE2, tryptase, MPO, adenosine) in NLF at specific time points compared to baseline | 0-21 days post challenge
Post LAIV change in overall "oxidative stress" in nasal epithelial cells | 0-21 days post challenge
Post LAIV change in epithelial gene expression profiles for innate immune and oxidant/antioxidant network arrays in nasal epithelial biopsies | 0-21 days post challenge
Change in levels and activities of circulating white blood cells, including eosinophils, basophils, monocytes, and lymphocytes | 0-21 days post challenge
Outcomes for GSTM1 null vs. sufficient genotype individuals | 0-21 days post challenge

CONTACTS AND LOCATIONS:
Overall Officials: Terry Noah, MD, Principal Investigator — University of North Carolina at Chapel Hill, Dept of Pediatrics / Center for Environmental Medicine, Asthma and Lung Biology
Locations (1):
- US EPA Human Studies Facility, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Pawlak EA, Noah TL, Zhou H, Chehrazi C, Robinette C, Diaz-Sanchez D, Muller L, Jaspers I. Diesel exposure suppresses natural killer cell function and resolution of eosinophil inflammation: a randomized controlled trial of exposure in allergic rhinitics. Part Fibre Toxicol. 2016 May 6;13(1):24. doi: 10.1186/s12989-016-0135-7. PMID 27154411
- [Derived] Noah TL, Zhou H, Zhang H, Horvath K, Robinette C, Kesic M, Meyer M, Diaz-Sanchez D, Jaspers I. Diesel exhaust exposure and nasal response to attenuated influenza in normal and allergic volunteers. Am J Respir Crit Care Med. 2012 Jan 15;185(2):179-85. doi: 10.1164/rccm.201103-0465OC. Epub 2011 Oct 27. PMID 22071326